CLINICAL TRIAL: NCT04365127
Title: A Single Center, Randomized, Controlled Trial of the Safety and Efficacy of Progesterone for the Treatment of COVID-19 in Hospitalized Men
Brief Title: Progesterone for the Treatment of COVID-19 in Hospitalized Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sara Ghandehari (Other)
Collaborators: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor-Investigator, Sara Ghandehari, Attending Physician, Internal Medicine/Pulmonary Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000611
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: COVID-19; Sars-CoV2
MeSH Terms: conditions — COVID-19 | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Progesterone plus SOC (Experimental): Progesterone 100 mg will be administered subcutaneously twice daily for 5 days in addition to institutional standard of care
  Interventions: Drug: Progesterone 100 MG
- SOC only (No Intervention): Subjects will receive institutional standard of care only

INTERVENTIONS:
Drug: Progesterone 100 MG — Subcutaneous administration twice daily
  Arms: Progesterone plus SOC

SUMMARY:
The purpose of this study is to assess safety and efficacy of progesterone for treatment of COVID-19 in hospitalized men.

DETAILED DESCRIPTION:
Hospitalized men with COVID-19 who meet the eligibility criteria will be informed about study and the potential risks. All the patients giving written informed consent will be randomized in 1:1 ratio to progesterone (100 mg SQ twice daily) plus standard of care or standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory-confirmed COVID-19 with in 72 hours prior to randomization
2. Respiratory symptoms or abnormal lung exam or abnormal chest imaging AND oxygen saturation ≤94% on room air, or requiring supplemental oxygen less than 50% high flow
3. Understands and agrees to comply with planned study procedures
4. Agrees to the collection of venous blood per protocol
5. Must agree to be placed on prophylactic dose of anticoagulation for prevention of deep venous thrombosis (DVT) while hospitalized

Exclusion Criteria:

1. ALT or AST >5 times the upper limit of normal
2. History of blood clots
3. History of breast cancer
4. Allergy to progesterone or betacyclodextrin
5. Use of supplemental oxygen prior to hospital admission
6. Requiring higher than 50% supplemental oxygen by high flow nasal cannula or mechanical ventilation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Change in clinical status of subjects at Day 7 based on the following 7-point ordinal scale | 7 days
  Change in clinical status of subjects at Day 7 based on the following 7-point ordinal scale
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen
  6. Not hospitalized, limitation on activities
  7. Not hospitalized, no limitations on activities

SECONDARY OUTCOMES:
Change in clinical status of subjects assessed daily while hospitalized and on Day 15 | 29 days
  Change in clinical status of subjects daily while hospitalized and at Day 15 based on the following 7-point ordinal scale
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen
  6. Not hospitalized, limitation on activities
  7. Not hospitalized, no limitations on activities
Duration of supplemental oxygen, mechanical ventilation (if applicable), and hospitalization | 15 days
  The length of time that the subjects require supplemental oxygen.
  The length of time that the subjects require mechanical ventilation (if applicable).
  The length of time that the subjects remain in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ghandehari, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Hall OJ, Klein SL. Progesterone-based compounds affect immune responses and susceptibility to infections at diverse mucosal sites. Mucosal Immunol. 2017 Sep;10(5):1097-1107. doi: 10.1038/mi.2017.35. Epub 2017 Apr 12. PMID 28401937
- [Background] Menzies FM, Henriquez FL, Alexander J, Roberts CW. Selective inhibition and augmentation of alternative macrophage activation by progesterone. Immunology. 2011 Nov;134(3):281-91. doi: 10.1111/j.1365-2567.2011.03488.x. PMID 21977998
- [Background] Jones LA, Anthony JP, Henriquez FL, Lyons RE, Nickdel MB, Carter KC, Alexander J, Roberts CW. Toll-like receptor-4-mediated macrophage activation is differentially regulated by progesterone via the glucocorticoid and progesterone receptors. Immunology. 2008 Sep;125(1):59-69. doi: 10.1111/j.1365-2567.2008.02820.x. Epub 2008 Mar 28. PMID 18373668
- [Background] Hall OJ, Limjunyawong N, Vermillion MS, Robinson DP, Wohlgemuth N, Pekosz A, Mitzner W, Klein SL. Progesterone-Based Therapy Protects Against Influenza by Promoting Lung Repair and Recovery in Females. PLoS Pathog. 2016 Sep 15;12(9):e1005840. doi: 10.1371/journal.ppat.1005840. eCollection 2016 Sep. PMID 27631986
- [Background] Breslin N, Baptiste C, Gyamfi-Bannerman C, Miller R, Martinez R, Bernstein K, Ring L, Landau R, Purisch S, Friedman AM, Fuchs K, Sutton D, Andrikopoulou M, Rupley D, Sheen JJ, Aubey J, Zork N, Moroz L, Mourad M, Wapner R, Simpson LL, D'Alton ME, Goffman D. Coronavirus disease 2019 infection among asymptomatic and symptomatic pregnant women: two weeks of confirmed presentations to an affiliated pair of New York City hospitals. Am J Obstet Gynecol MFM. 2020 May;2(2):100118. doi: 10.1016/j.ajogmf.2020.100118. Epub 2020 Apr 9. PMID 32292903
- [Background] Cometti B. Pharmaceutical and clinical development of a novel progesterone formulation. Acta Obstet Gynecol Scand. 2015 Nov;94 Suppl 161:28-37. doi: 10.1111/aogs.12765. PMID 26342177
- [Background] Doblinger J, Cometti B, Trevisan S, Griesinger G. Subcutaneous Progesterone Is Effective and Safe for Luteal Phase Support in IVF: An Individual Patient Data Meta-Analysis of the Phase III Trials. PLoS One. 2016 Mar 18;11(3):e0151388. doi: 10.1371/journal.pone.0151388. eCollection 2016. PMID 26991890
- [Background] Chen T, Wu D, Chen H, Yan W, Yang D, Chen G, Ma K, Xu D, Yu H, Wang H, Wang T, Guo W, Chen J, Ding C, Zhang X, Huang J, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical characteristics of 113 deceased patients with coronavirus disease 2019: retrospective study. BMJ. 2020 Mar 26;368:m1091. doi: 10.1136/bmj.m1091. PMID 32217556
- [Derived] Ghandehari S, Matusov Y, Pepkowitz S, Stein D, Kaderi T, Narayanan D, Hwang J, Chang S, Goodman R, Ghandehari H, Mirocha J, Bresee C, Tapson V, Lewis M. Progesterone in Addition to Standard of Care vs Standard of Care Alone in the Treatment of Men Hospitalized With Moderate to Severe COVID-19: A Randomized, Controlled Pilot Trial. Chest. 2021 Jul;160(1):74-84. doi: 10.1016/j.chest.2021.02.024. Epub 2021 Feb 20. PMID 33621601